CLINICAL TRIAL: NCT04953650
Title: The Effectiveness of Intermittent Fasting Towards Elevated Blood Pressure Among Civil Servants in Aceh
Brief Title: Intermittent Fasting Towards Elevated Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Collaborators: University of Muhammadiyah Aceh (Other)
Responsible Party: Principal Investigator, Mas Ayu binti Said, Academician, University of Malaya
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Intermittent Fasting
Record Dates: First submitted 2021-06-15; First posted 2021-07-08 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Intermittent Fasting; Elevated Blood Pressure
Keywords: fasting; intermittent fasting; 5:2 diet; blood pressure; body mass index; body weight; waist circummference; calorie intake
MeSH Terms: conditions — Intermittent Fasting; Hypertension; Fasting; Body Weight

STUDY DESIGN:
Intervention Model Description: This trial will have two groups; the intervention and the control group. Both groups will receive health education. Hence, the Intervention group will undergo two fasting days within the week from dusk to dawn, while the control group is doing the regular diet. No exercise control for both groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): two fasting days and five ad-libitum days followed by usual exercise.
  Interventions: Behavioral: Intermittent fasting
- Control group (Sham Comparator): Usual diet and usual exercise prior to the intervention.
  Interventions: Other: No intervention

INTERVENTIONS:
Behavioral: Intermittent fasting — The intervention group is required to perform intermittent fasting for two days. The intermittent fasting method for this group will mimic the Sunnah Muslim fasting; they are allowed to consume food and calorie water without restriction in between dusk and dawn. During the five ad libitum days, they are allowed to have a variety of foods and drinks. Subjects will be informed about healthy food choices; choosing low-fat meat and dairy options, increasing fruit and vegetable intake.
  Arms: intervention group
Other: No intervention — The control group will receive education training at the baseline as well, regarding blood pressure and nutrition. They will have usual exercise prior to the intervention. Furthermore, the group will have equal health education through health promotion leaflets which have been issued by the ministry of health.
  Arms: Control group

SUMMARY:
To date, the prevalence of Hypertension (HPT) is getting increase worldwide. This situation is contributed mostly by the Lower-Income Countries (LIC) and Lower-Middle-Income Countries (LMICs) include Asians. Elevated Blood Pressure (EBP) in the early phase is often unrealized before developing to HPT, leading to several diseases in terms of cardiovascular diseases (CVDs). In preventing EBP, the European Society of Cardiology in 2017 classifies blood pressure into three groups; normal, pre-hypertension, and hypertensive crisis. People in the normal phase with the high-normal line are classified into EBP. If this group is determined and controlled, they will further keep in normal blood pressure. Contrarily, they are experiencing the next phase of HPT.

Like other Asian countries, Indonesia was experiencing an extreme prevalence of HPT, and Aceh, which is one of the provinces in Indonesia has a very high prevalence of HPT as well (20% increment from 2013-2018), is estimated to equal to the EBP prevalence. Despite many promotive and preventive interventions confirmed to decrease HPT, early screening has been convinced to recover the HPT in Indonesia. However, the HPT prevalence was examined steadily increasing. Intermittent fasting (IF) is recognized as a new method in decreasing metabolic factors based on several types of research currently. Therefore, the investigators are studying the effectiveness of intermittent fasting on people with EBP. Conducting healthy lifestyle intervention that is inexpensive, doable, and easily accessible, would be a new method for controlling EBP.

DETAILED DESCRIPTION:
This trial aims to evaluate the effectiveness of three months intermittent fasting intervention followed by three months maintenance phase in stabilizing blood pressure among the EBP group with the high-normal signal. This trial will conducts in Aceh, Indonesia.

Trial procedure

1. In the beginning, the researcher chooses the allocation group for either intervention or control group based on the potential number of workers from each department. Based on that, it was decided that the intervention group is the Governor's office, and the Aceh Besar regency secretariat is the control group.
2. Letters of permission are submitted to both departments and continued by blood pressure screening once it is approved. Hence, the enumerators will screen all the workers. Each eligible participant (EBP 130-139/85-89 mm Hg and BMI ³ 25 kilograms/m2) will be invited to join blood pressure plus nutrition class on the day after, and fulfill the baseline characteristic questionnaire once they sign the informed consent. During the class, the researcher will describe the study procedure, study objective, process, monitoring, follow-up, methodology, risk and benefit, confidentiality, anonymity, and withdrawal from the study in both groups with the different context of intervention. Because of the covid-19 pandemic, all participants are allocated in a few small groups during baseline training.
3. The participants will join complete anthropometric measurements and fulfill questions in the STEP instrument and GPAQ instrument. Four enumerators will assist the participants; however, they will be blinded to intervention assignment.
4. The intervention group will undergo two fasting days and five ad libitum days during the intervention phase and continued to the maintenance phase. Otherwise, the control group will have a usual diet before the trial. Furthermore, both groups will have current exercise.
5. Calculation of the actual sample size to detect effect size in the primary and secondary objectives of the project has been conducted. Sample selection techniques will be described further in the published paper.
6. A mixed linear model will be applied to count the intervention effects (blood pressure, body weight, body mass index, waist circumference, and calorie intake), while a generalized estimating equation (GEE) will be used as well for categorical outcomes. Characteristics at baseline will be summarised by each arm using numbers and percentages, means and standard deviations or medians, and inter-quartile ranges where applicable.

ELIGIBILITY:
Inclusion Criteria:

1. Adult between 18-60 years with EBP 130-139/85-89 mm Hg;
2. Overweight and obese with BMI above is equal to 25 kilogram/m2;
3. Do not have any gastric diseases or problems with the fasting;
4. Able to read and write;
5. Willing to sign the inform consent

Exclusion Criteria:

1. Disability person;
2. In medication either blood pressure or another disease;
3. Pregnant woman;
4. Employees who will be retired in the intervention duration;
5. Employees who will undergo hajj pilgrimage in the year 2021.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2022-03-13 (Actual); Study Completion 2022-03-13 (Actual)

PRIMARY OUTCOMES:
Blood pressure | Baseline, 12 weeks and 24 weeks
  Change from baseline systolic blood pressure and diastolic blood pressure at 12 weeks and 24 weeks (6 months) in participants with elevated blood pressure and BMI above is equal to 25 kilogram/m2.
  The blood pressure is measured by Omron sphygmomanometer (Omron HEM 7130 LP, Kyoto, Japan).

SECONDARY OUTCOMES:
Body weight | Baseline, 12 weeks and 24 weeks
  Change from baseline body weight at 12 weeks and 24 weeks (6 months) in participants with elevated blood pressure and BMI above is equal to 25 kilogram/m2.
  The body weight is measured by weighing scale (Oserio Body fat monitor, Guozhong, Taiwan)
Body mass index | Baseline, 12 weeks and 24 weeks
  Change from baseline BMI at 12 weeks and 24 weeks (6 months) in participants with elevated blood pressure and BMI above is equal to 25 kilogram/m2.
  The BMI is measured by weighing scale (Oserio Body fat monitor, Guozhong, Taiwan) and Stadiometer (Saga, Indonesia)
Waist circumference | Baseline, 12 weeks and 24 weeks
  Change from baseline waist circumference at 12 weeks and 24 weeks (6 months) in participants with elevated blood pressure and BMI above is equal to 25 kilogram/m2.
  The waist circumference is measured by tape line (China)
Calorie intake | Baseline, 12 weeks and 24 weeks
  Change from baseline calorie intake at 12 weeks and 24 weeks (6 months) in participants with elevated blood pressure and BMI above is equal to 25 kilogram/m2.
  The calorie intake is measured by three days food record form.

CONTACTS AND LOCATIONS:
Overall Officials: Mas Ayu Said, MPH, PhD, Principal Investigator — University of Malaya
Locations (1):
- Aceh Governor's Office and Aceh Besar regency secretariat, Banda Aceh, Special Region of Aceh, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allaert FA. Effect of NaCl + Chitosan 3% vs. NaCl on high blood pressure parameters of healthy volunteers with prehypertension. Minerva Cardioangiol. 2017 Dec;65(6):563-576. doi: 10.23736/S0026-4725.17.04451-6. Epub 2017 Aug 31. PMID 28862406
- [Background] Irwan AM, Kato M, Kitaoka K, Ueno E, Tsujiguchi H, Shogenji M. Development of the salt-reduction and efficacy-maintenance program in Indonesia. Nurs Health Sci. 2016 Dec;18(4):519-532. doi: 10.1111/nhs.12305. Epub 2016 Sep 29. PMID 27687887
- [Background] Jamshed H, Beyl RA, Della Manna DL, Yang ES, Ravussin E, Peterson CM. Early Time-Restricted Feeding Improves 24-Hour Glucose Levels and Affects Markers of the Circadian Clock, Aging, and Autophagy in Humans. Nutrients. 2019 May 30;11(6):1234. doi: 10.3390/nu11061234. PMID 31151228
- [Background] Hoddy KK, Kroeger CM, Trepanowski JF, Barnosky A, Bhutani S, Varady KA. Meal timing during alternate day fasting: Impact on body weight and cardiovascular disease risk in obese adults. Obesity (Silver Spring). 2014 Dec;22(12):2524-31. doi: 10.1002/oby.20909. Epub 2014 Sep 24. PMID 25251676
- [Background] Kerr DA, Dhaliwal SS, Pollard CM, Norman R, Wright JL, Harray AJ, Shoneye CL, Solah VA, Hunt WJ, Zhu F, Delp EJ, Boushey CJ. BMI is Associated with the Willingness to Record Diet with a Mobile Food Record among Adults Participating in Dietary Interventions. Nutrients. 2017 Mar 7;9(3):244. doi: 10.3390/nu9030244. PMID 28272343
- [Background] Kusuma D, Kusumawardani N, Ahsan A, K Sebayang S, Amir V, Ng N. On the verge of a chronic disease epidemic: comprehensive policies and actions are needed in Indonesia. Int Health. 2019 Nov 13;11(6):422-424. doi: 10.1093/inthealth/ihz025. PMID 31294789
- [Background] Bowen J, Brindal E, James-Martin G, Noakes M. Randomized Trial of a High Protein, Partial Meal Replacement Program with or without Alternate Day Fasting: Similar Effects on Weight Loss, Retention Status, Nutritional, Metabolic, and Behavioral Outcomes. Nutrients. 2018 Aug 23;10(9):1145. doi: 10.3390/nu10091145. PMID 30142886
- [Result] Whelton PK, Carey RM, Aronow WS, Casey DE Jr, Collins KJ, Dennison Himmelfarb C, DePalma SM, Gidding S, Jamerson KA, Jones DW, MacLaughlin EJ, Muntner P, Ovbiagele B, Smith SC Jr, Spencer CC, Stafford RS, Taler SJ, Thomas RJ, Williams KA Sr, Williamson JD, Wright JT Jr. 2017 ACC/AHA/AAPA/ABC/ACPM/AGS/APhA/ASH/ASPC/NMA/PCNA Guideline for the Prevention, Detection, Evaluation, and Management of High Blood Pressure in Adults: Executive Summary: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Circulation. 2018 Oct 23;138(17):e426-e483. doi: 10.1161/CIR.0000000000000597. No abstract available. PMID 30354655
- [Result] Sutton EF, Beyl R, Early KS, Cefalu WT, Ravussin E, Peterson CM. Early Time-Restricted Feeding Improves Insulin Sensitivity, Blood Pressure, and Oxidative Stress Even without Weight Loss in Men with Prediabetes. Cell Metab. 2018 Jun 5;27(6):1212-1221.e3. doi: 10.1016/j.cmet.2018.04.010. Epub 2018 May 10. PMID 29754952
- [Result] Sundfor TM, Svendsen M, Tonstad S. Effect of intermittent versus continuous energy restriction on weight loss, maintenance and cardiometabolic risk: A randomized 1-year trial. Nutr Metab Cardiovasc Dis. 2018 Jul;28(7):698-706. doi: 10.1016/j.numecd.2018.03.009. Epub 2018 Mar 29. PMID 29778565
- [Result] Bhutani S, Klempel MC, Kroeger CM, Trepanowski JF, Varady KA. Alternate day fasting and endurance exercise combine to reduce body weight and favorably alter plasma lipids in obese humans. Obesity (Silver Spring). 2013 Jul;21(7):1370-9. doi: 10.1002/oby.20353. Epub 2013 May 29. PMID 23408502
- [Derived] Baharuddin D, Said MA, Majid HA. Protocol For Intervention Study In Reducing Elevated Blood Pressure Through Intermittent Fasting. J Pak Med Assoc. 2023 Nov;73(11):2171-2176. doi: 10.47391/JPMA.7748. PMID 38013523